CLINICAL TRIAL: NCT01110889
Title: An 8-week, Randomized, Double-blind, Placebo-controlled, Parallel-group, Multi-center Study of the Efficacy and Safety of Agomelatine 0.5 mg and 1 mg Sublingual Tablets Administered Once Daily in Patients With Major Depressive Disorder (MDD)
Brief Title: Efficacy, Safety and Tolerability of Agomelatine Sublingual Tablets in the Treatment of Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAGO178C2301
Record Dates: First submitted 2010-04-23; First posted 2010-04-27 (Estimated); Last update posted 2020-12-23 (Actual); Status verified 2013-02

CONDITIONS: Major Depressive Disorder
Keywords: Agomelatine; Major Depressive Disorder; MDD; depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — agomelatine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- AGO178C 0.5 mg /day (Experimental)
  Interventions: Drug: Agomelatine (AGO178C)
- AGO178C 1 mg / day (Experimental)
  Interventions: Drug: Agomelatine (AGO178C)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Agomelatine (AGO178C)
  Arms: AGO178C 0.5 mg /day
Drug: Agomelatine (AGO178C)
  Arms: AGO178C 1 mg / day
Drug: Placebo
  Arms: Placebo

SUMMARY:
The study will assess efficacy, safety and tolerability of 0.5 mg/day and 1 mg/day of sublingual (under the tongue) formulation of agomelatine in patients with Major Depressive Disorder. This study includes an 8-week double-blind phase.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of MDD, single or recurrent episode, according to DSM-IV criteria.
* Current episode ≥4 weeks.
* CGI-Severity score ≥4 at Screening and Baseline.

Exclusion Criteria:

* History of bipolar disorder (I or II), schizophrenia, schizoaffective disorder, eating disorder (current or during previous one year), obsessive-compulsive disorder.
* Any other current Axis I disorder other than MDD which is the focus of treatment.
* Substance or alcohol abuse in the last 30 days, dependence in the last 6 months.
* Concomitant psychotropic medication, including herbal preparations and melatonin.
* Psychotherapy of any type.
* Prior exposure to agomelatine.
* Female patients of childbearing potential who are not using effective contraception.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 582 (Actual)
Dates: Start 2010-05; Primary Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Change from Baseline to endpoint at Week 8 using the total score of the Hamilton Depression Rating Scale | Baseline and 8 weeks

SECONDARY OUTCOMES:
Effect on subjective sleep, as measured by the score of the Leeds Sleep Evaluation Questionnaire (LSEQ) domain "quality of sleep" at Week 8 | 8 weeks
Proportion of patients who demonstrate clinical response, where response is defined by a reduction of at least 50% in the Baseline clinician-rated HAM-D total score at Week 8 endpoint | 8 weeks
Proportion of patients who demonstrate clinical improvement at Week 8, where improvement is defined by a score of 1 or 2 on the CGI-I scale | 8 weeks
Proportion of patients who achieve remission | 8 weeks
Safety and tolerability by adverse events and serious adverse events, and assessment of suicidal ideation and behavior by Columbia Suicide Severity Rating Scale. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (48):
- United States (47):
  - Birmingham Psychiatry, Birmingham, Alabama
  - Southwestern Research Institute, Beverly Hills, California
  - Pharmacology Research Institute, Encino, California
  - Mood & Anxiety Research, Fresno, California
  - Excell Research, Inc, Oceanside, California
  - Cnri-La, Llc, Pico Rivera, California
  - CNRI San Diego, San Diego, California
  - University of California San Diego Medical Center, San Diego, California
  - University of Colorado Denver, Aurora, Colorado
  - Western Affiliated Research Institute, Denver, Colorado
  - Clinical Research Institute of South Florida, Hialeah, Florida
  - Florida Clinical Research Center LLC, Maitland, Florida
  - CNS Healthcare, Orlando, Florida
  - Broward Research Group, Pembroke Pines, Florida
  - Quantum Lab. N. Broward Memory Disorder Center, Pompano Beach, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Northwest Behavioral Research Center, Marietta, Georgia
  - Hawaii Clinical Research Center, Honolulu, Hawaii
  - Mountain West Clinical Trials, Eagle, Idaho
  - Rush University Medical Center, Chicago, Illinois
  - Psychiatric Associates, Overland Park, Kansas
  - CTT Clinical Trials Technology, Prairie Village, Kansas
  - Clinical Trials Management, Metairie, Louisiana
  - Mount Auburn Medical Associates, Watertown, Massachusetts
  - Coastal Research Associates, Weymouth, Massachusetts
  - Comprehensive Psychiatric Associates, Gladstone, Missouri
  - Psychopharmacology Research Association of Princeton, Princeton, New Jersey
  - Bio Behavioral Health, Toms River, New Jersey
  - Albuquerque Neuroscience, Albuquerque, New Mexico
  - Neurological Associates Of Albany, P.C., Albany, New York
  - Neurobehavioral Research Inc., Cedarhurst, New York
  - Finger Lakes Clinical Research, Rochester, New York
  - Montefiore Medical Center, The Bronx, New York
  - Odyssey Research Services, Fargo, North Dakota
  - The Ohio State University - Harding Hospital, Columbus, Ohio
  - Midwest Clinical Research Center, Dayton, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Cutting Edge Research, Oklahoma City, Oklahoma
  - Sunstone Medical Research, LLC, Medford, Oregon
  - Lehigh Center for Clinical Research, Allentown, Pennsylvania
  - Psychiatric Consultants, Franklin, Tennessee
  - KRK Medical Research, Dallas, Texas
  - FutureSearch Trials of Dallas, Dallas, Texas
  - InSite Clinical Research, DeSoto, Texas
  - Texas Center for Drug Development, Houston, Texas
  - Alliance Research Group, LLC, Richmond, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
- Inspira Clinical Research, San Juan, Puerto Rico

REFERENCES:
- See also: https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=6663 — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=6563